CLINICAL TRIAL: NCT04851249
Title: Hallux Valgus - Radiological and Clinical Predictors for Outcome After Surgery
Brief Title: Hallux Valgus- Radiological and Clinical Predictors for Outcome After Surgery
Status: Recruiting | Type: Observational
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 217200
Record Dates: First submitted 2021-04-09; First posted 2021-04-20 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Hallux Valgus
Keywords: Hallux valgus; Outcome predictors; MOXFQ
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult participants operated for Hallux Valgus deformity: All adult participants accepted for hallux valgus corrective surgery at ostfold hospital trust (ØHT) is asked to participate in the study. The goal is to include 200-250 participants.
  Interventions: Procedure: Hallux Valgus - chevron osteotomy, lapidus procedure

INTERVENTIONS:
Procedure: Hallux Valgus - chevron osteotomy, lapidus procedure — The purpose is to compare the preoperative clinical features (previous medical history, age, BMI, occupational status etc), PROMs (Manchester-Oxford Foot and ankle questionnaire, SF-36, VAS activity scale) and radiological parameters (both two and three dimensional) with the postoperative PROMs (+ likert scale) and the postoperative radiological parameters.

SUMMARY:
Prospective observational study to evaluate the clinical and radiological predictors for outcome in hallux valgus (HV) corrective surgery.

DETAILED DESCRIPTION:
Hallux valgus (HV) is the most common deformity in the adult forefoot. Characterizing and classifying HV primarily has been based on weightbearing radiographic imaging. Understanding of this pathologic process has mainly been confined to two planes, where the dominating modality of choice has been assessment by antero-posterior (AP) and lateral radiographs. From these two projections, imaging parameters have developed to define the severity of HV. With this understanding as the basis for describing the deformity, more than 140 operative techniques have been described. Although many of these techniques are of historical interest only, consistently favourable outcomes remain elusive even among more popular current techniques. HV corrective surgery is known to have mediocre results, with recurrence rate as high as 30-70%. Unsuccessful treatment of the condition is amongst the most common in the Norwegian patient injury compensation scheme. The variation in corrective techniques and the associated persistent and clinically significant rates of poor outcomes may indicate an incomplete treatment of the pathoanatomy of HV. Numerous recent publications have proved that the hallux valgus deformity should be viewed as a three-dimensional deformity. These recent studies have also pointed out new radiological parameters in AP and axial view, focusing on the multiplanar understanding of the deformity. The key challenge of the hallux valgus foot is the lack of clear guidelines for choosing the best treatment to these large group of patients. There is of today no guidelines nor consensus considering the indication for surgical treatment of the hallux valgus deformity. It is not known how much nuisance the patient should present before surgery could be worthwhile. Many studies have been made in the field of HV, but literature with the focus on comparing the surgical correction and the patient related clinical outcome is sparse and insufficient.

In this project the investigators primary aim is to investigate radiological and clinical factors that predict outcome in participants operated for hallux valgus deformity.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients accepted for hallux valgus surgery (mild, moderate, severe) at the ØHT will be asked to participate in the study

Exclusion Criteria:

* Previous hallux valgus surgery in the same foot
* Lack of compliance
* Not available for follow-up
* Language difficulties (not able to communicate in English or Norwegian)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients accepted for hallux valgus surgery at the ØHT
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparing the pre and postoperative Manchester-Oxford Foot Questionnaire (MOXFQ) index score in participants operated for hallux valgus deformity | Participant enrollment is expected to be completed within 3-4 years time, they will be evaluated preoperatively, 6 weeks, 12 weeks and 52 weeks postoperatively
  The MOXFQ (Dawson et al., 2006) was developed to measure perceived foot-specific functioning and health-related quality of life. The MOXFQ is supported as the current most valid, reliable and responsive foot & ankle instrument (Jia, Huang&Gagnier, 2017). It is available in Norwegian, but has not been validated in its translated form. The score compromises a total of 16 items. They are distributed within 3 dimensions; foot pain (5 items), walking/standing (7 items) and social interaction (4 items) where all items are scored on a 5-point Likert scale, score 0 (best) to 4 (worst). The MOXFQ index score (Morely et al., 2013) will be used as the main outcome and we define an increase of at least 15 points as a successful outcome. We plan to run multiple regression analysis with baseline parameters as well as radiological and Patient-reported outcome measures (PROMs) data as predictors. To account for loss to follow-up we will include 250 patients in this study.

SECONDARY OUTCOMES:
Comparing the traditional and newer rotational radiological parameters with PROMs pre and postoperatively | Participant enrollment is expected to be completed within 3-4 years time, patient follow-up 6, 12 and 52 weeks postoperatively. Goal of inclusion 250 patients.
  Investing the correlation between the traditional and newer rotational parameters on weighted anterior-posterior and axial radiograph of the forefoot (lateral head shape of first metatarsal, hardy and Clapham tibial sesamoid position, joint congruity, distal metatarsal articular angle (DMAA), intermetatarsal angle (IMA), hallux valgus angle (HVA), metatarsal rotational angle, sesamoid rotational angle) and the PROMs (MOxFQ, SF-36, visual analogue scale (VAS) activity, likert scale) pre and postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Marius Molund, MD, PhD, Study Director — Head of foot and ankle department at ØHT
Locations (1):
- Østfold Hospital Trust, Sarpsborg, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: Undecided